CLINICAL TRIAL: NCT03369236
Title: A Phase 2, Proof-of-Concept, Randomized, Double-Blinded, Placebo-Controlled Study of ACH-0144471 Treatment for 6 Months in Patients With C3 Glomerulopathy (C3G), With an Open-label Extension
Brief Title: A Proof-of-Concept Study of Danicopan for 6 Months of Treatment in Participants With C3 Glomerulopathy (C3G)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH471-204; 2017-000663-33 (EudraCT Number)
Record Dates: First submitted 2017-11-17; First posted 2017-12-11 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: C3 Glomerulopathy; C3 Glomerulonephritis; Dense Deposit Disease
Keywords: factor D; fD; Alternative pathway; Complement mediated disease; Membranoproliferative Glomerulonephritis; Primary MPGN; MPGN; Mesangiocapillary Glomerulonephritis; Idiopathic MPGN; DDD; C3GN
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigator and participant blinded; Sponsor open. Participants were randomized 1:1 to receive either danicopan or placebo for a period of 6 months, followed by an open-label extension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Danicopan (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period) (Active Comparator): Danicopan was administered at a starting dose of 100 milligrams (mg) 3 times daily (TID) for the first 2 weeks, then dosage was to be increased to 200 mg TID for the remainder of the 6-month treatment period.
  All participants who completed the double-blind treatment period were enrolled in the open-label extension period and were to receive danicopan 200 mg TID.
  Interventions: Drug: Danicopan
- Placebo (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period) (Placebo Comparator): Placebo was administered TID during the 6-month treatment period.
  All participants who completed the double-blind treatment period were enrolled in the open-label extension period and were to receive danicopan 200 mg TID.
  Interventions: Drug: Danicopan; Drug: Placebo

INTERVENTIONS:
Drug: Danicopan — Danicopan was administered as an oral tablet.
  Other Names: ACH-4471; ACH4471; 4471; ACH-0144471 (formerly); ALXN2040
Drug: Placebo — Matching placebo was administered as an oral tablet.
  Arms: Placebo (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period)

SUMMARY:
The primary purpose of this proof-of-concept clinical study was to evaluate the efficacy and safety of the study drug, ACH-0144471 (also known as danicopan and ALXN2040), in participants with C3G who also had significant proteinuria attributable to C3G.

ELIGIBILITY:
Key Inclusion Criteria:

* Had biopsy-confirmed primary C3G
* Had clinical evidence of ongoing disease based on significant proteinuria, attributable to C3G disease in the opinion of the Principal Investigator (PI), and present prior to study entry and confirmed during Screening
* Was willing to comply with vaccination requirements.

Key Exclusion Criteria:

* Had a history or presence of any clinically relevant co-morbidities that would make the participant inappropriate for the study
* Had ever received danicopan
* Had more than 50% fibrosis or more than 50% of glomeruli with cellular crescents on the pre-treatment renal biopsy
* Had an estimated glomerular filtration rate <30 milliliters/minute/1.73 meters squared at the time of screening or at any time over the preceding 4 weeks
* Was a renal transplant recipient or receiving renal replacement therapy
* Had a history of a major organ transplant or hematopoietic stem cell/marrow transplant
* Had evidence of monoclonal gammopathy of unclear significance, infections, malignancy, autoimmune diseases, or other conditions to which C3G is secondary
* Had other renal diseases that would interfere with interpretation of the study
* Had been diagnosed with or showed evidence of hepatobiliary cholestasis
* Females who were pregnant, nursing, or planning to become pregnant during the study or within 90 days of study drug administration
* Had a history of febrile illness, a body temperature >38°Celsius, or other evidence of a clinically significant active infection, within 14 days prior to study drug administration
* Had evidence of human immunodeficiency virus, hepatitis B infection, or active hepatitis C infection at Screening
* Had laboratory abnormalities at screening that, in the opinion of the PI, would make the participant inappropriate for the study

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Clinical Study Site, Aurora, Colorado
  - Clinical Study Site, Lawrenceville, Georgia
  - Clinical Study Site, Iowa City, Iowa
  - Clinical Study Site, Baltimore, Maryland
  - Clinical Study Site, New York, New York
- Clinical Study Site, London, United Kingdom

REFERENCES:
- [Derived] Nester C, Appel GB, Bomback AS, Bouman KP, Cook HT, Daina E, Dixon BP, Rice K, Najafian N, Hui J, Podos SD, Langman CB, Lightstone L, Parikh SV, Pickering MC, Sperati CJ, Trachtman H, Tumlin J, de Vries AP, Wetzels JFM, Remuzzi G. Clinical Outcomes of Patients with C3G or IC-MPGN Treated with the Factor D Inhibitor Danicopan: Final Results from Two Phase 2 Studies. Am J Nephrol. 2022;53(10):687-700. doi: 10.1159/000527167. Epub 2022 Nov 24. PMID 36423588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To enroll in the study, participants were required to have a biopsy confirmed diagnosis of C3 Glomerulopathy (C3G), with initial diagnosis made at least 3 months prior to dosing and significant proteinuria.
Period: Double-blind Treatment Period
Arm/Group | Danicopan (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period) | Placebo (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period)
Started | 6 | 7
Received at Least 1 Dose of Study Drug | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Accidental unblinding | 0 | 1
Period: Open-label Extension Period
Arm/Group | Danicopan (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period) | Placebo (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period)
Started | 6 | 6
Received at Least 1 Dose of Study Drug | 6 (All participants received danicopan in the open-label extension period.) | 6 (All participants received danicopan in the open-label extension period.)
Completed | 1 | 0
Not Completed | 5 | 6
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Sponsor decision to close study | 3 | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug during the double-blind treatment period.
Groups:
- Danicopan (Double-blind Treatment Period): Danicopan was administered at a starting dose of 100 mg 3 times daily (TID) for the first 2 weeks, then dosage was to be increased to 200 mg TID for the remainder of the 6-month treatment period.
- Placebo (Double-blind Treatment Period): Placebo was administered TID during the 6-month treatment period.
- Total: Total of all reporting groups
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period) | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (10.54) | 24.9 (4.85) | 25.2 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 2
  White | 5 | 4 | 9
  Other | 1 | 1 | 2
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
  United Kingdom | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Composite Biopsy Score At Week 28
Description: The composite biopsy score was based on a score incorporating changes in the activity index, glomerular C3c staining, and glomerular macrophage infiltration at the end of 6 months of treatment. The composite renal biopsy index scoring system ranged from 0 to 21, with higher scores indicating worse outcomes.
Time Frame: Baseline, Week 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Danicopan (Double-blind Treatment Period): Danicopan was administered at a starting dose of 100 mg TID for the first 2 weeks, then dosage was to be increased to 200 mg TID for the remainder of the 6-month treatment period.
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 11.7 (4.23) | 9.3 (3.50)
  Week 28: number analyzed (Participants) | 6 | 5
  Week 28 | 9.2 (4.87) | 10.7 (3.39)
  Change from Baseline: number analyzed (Participants) | 6 | 5
  Change from Baseline | -2.0 (1.87) | 1.3 (2.88)

2. Primary Outcome: Participants With Reduction In Proteinuria At Week 28
Description: Proteinuria reduction was defined as ≥ 30% decrease from baseline based on 24-hour urine protein (mg/day).
Time Frame: Week 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Number; unit: participants
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
Number analyzed (Participants) | 4 | 5
participants | 0 | 1

3. Secondary Outcome: Change From Baseline In Proteinuria At Week 28
Description: Proteinuria was assessed based on 24-hour urine collections at baseline and Week 28.
Time Frame: Baseline, Week 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
Number analyzed (Participants) | 6 | 7
mg/day
  Baseline | 6137.67 (2904.359) | 4274.47 (2992.819)
  Week 28: number analyzed (Participants) | 4 | 5
  Week 28 | 5301.75 (2984.445) | 5186.80 (4069.279)
  Change from Baseline: number analyzed (Participants) | 4 | 5
  Change from Baseline | 302.00 (764.211) | 182.20 (994.558)

4. Secondary Outcome: Percent Change From Baseline In Proteinuria At Week 28
Description: Proteinuria was assessed based on 24-hour urine collections at baseline and Week 28.
Time Frame: Baseline, Week 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
Number analyzed (Participants) | 4 | 5
percent change | 12.5 (31.11) | -10.4 (31.35)

5. Secondary Outcome: Slope Of Estimated Glomerular Filtration Rate (eGFR) From Baseline To 6 Months
Description: Slope of eGFR was estimated using a simple linear regression for each participant, including all data values from baseline until the end of the 6-month blinded treatment period, with eGFR as the dependent variable and time as the independent variable.
Time Frame: 6 months
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2 per month
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
Number analyzed (Participants) | 6 | 7
mL/min/1.73 m^2 per month | -2.26840 (1.790814) | -1.45421 (2.228395)

6. Secondary Outcome: Slope Of Estimated Glomerular Filtration Rate (eGFR) After Open-label Danicopan Treatment
Description: Slope of eGFR was estimated using a simple linear regression for each participant, including all data values during the open-label extension period with eGFR as the dependent variable and time as the independent variable.
Time Frame: 12 months
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2 per month
Groups:
- Danicopan (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period: Danicopan was administered at a starting dose of 100 mg TID for the first 2 weeks, then dosage was to be increased to 200 mg TID for the remainder of the 6-month treatment period.
  All participants who completed the double-blind treatment period were enrolled in the open-label extension period and were to receive danicopan 200 mg TID.
- Total: All participants who received danicopan or placebo during the 6-month treatment period followed by danicopan 200 mg TID in the extension period.
Arm/Group | Danicopan (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period | Placebo (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period) | Total
Number analyzed (Participants) | 5 | 4 | 9
mL/min/1.73 m^2 per month | -1.02556 (1.389128) | -1.84935 (3.506810) | -1.39169 (2.401039)

7. Secondary Outcome: Change From Baseline In eGFR At Week 28
Description: Change from baseline in eGFR at Week 28 is presented.
Time Frame: Baseline, Week 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
Number analyzed (Participants) | 6 | 7
mL/min/1.73 m^2
  Baseline | 79.890 (44.4571) | 68.381 (36.7249)
  Week 28: number analyzed (Participants) | 6 | 5
  Week 28 | 67.543 (47.8062) | 50.874 (15.0517)
  Change from Baseline: number analyzed (Participants) | 6 | 5
  Change from Baseline | -12.347 (10.8063) | -8.700 (16.0990)

8. Secondary Outcome: Participants With Significant Improvement In eGFR Relative To Baseline At Week 28
Description: Significant improvement relative to baseline was defined as a ≥ 20% increase from baseline in eGFR.
Time Frame: Baseline, Week 28
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Number; unit: participants
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
Number analyzed (Participants) | 6 | 5
participants | 0 | 0

9. Secondary Outcome: Participants With Significant Improvement In eGFR Relative To Baseline At Week 52
Description: Significant improvement relative to baseline was defined as a ≥ 20% increase from baseline in eGFR.
Time Frame: Baseline, Week 52
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Number; unit: participants
Groups:
- Danicopan (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period): Danicopan was administered at a starting dose of 100 mg TID for the first 2 weeks, then dosage was to be increased to 200 mg TID for the remainder of the 6-month treatment period.
  All participants who completed the double-blind treatment period were enrolled in the open-label extension period and were to receive danicopan 200 mg TID.
Arm/Group | Danicopan (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period) | Placebo (Double-blind Treatment Period), Followed by Danicopan (Open-label Extension Period)
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Week 28 (treatment period and follow-up) and Week 104 (open-label extension and follow-up). The median study duration was 548.0 days.
Groups:
- Danicopan (Open-label Extension Period): All participants who received danicopan or placebo in the treatment period were to receive danicopan 200 mg TID during the open-label extension period.
Arm/Group | Danicopan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period) | Danicopan (Open-label Extension Period)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 1/12
Other Adverse Events (participants affected / at risk) | 5/6 | 5/7 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danicopan (Double-blind Treatment Period) (N=6) | Placebo (Double-blind Treatment Period) (N=7) | Danicopan (Open-label Extension Period) (N=12)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danicopan (Double-blind Treatment Period) (N=6) | Placebo (Double-blind Treatment Period) (N=7) | Danicopan (Open-label Extension Period) (N=12)
Haematoma (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0
Pregnancy of partner (Social circumstances) | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Dizziness (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03369236/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT03369236/SAP_001.pdf